CLINICAL TRIAL: NCT01762787
Title: A Randomised, Single Blind, Placebo-Controlled, Cross-over, Phase 1 Methodology Study to Validate the Cantharidin Blister Model in Healthy Male Volunteers
Brief Title: Phase I Methodology Study to Validate the Cantharidin Blister Model in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 114416
Record Dates: First submitted 2012-11-28; First posted 2013-01-08 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Aspirin; Prednisolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Effect of Aspirin (Active Comparator): Positive control as previously used in the cantharidin blister experimental model of inflammation
  Interventions: Drug: Cantharidin solution; Drug: Aspirin; Drug: Placebo to aspirin
- Effect of steroid - Prednisolone (Experimental): Prednisolone selected as steroids should provide the most robust positive control anti-inflammatory therapy
  Interventions: Drug: Cantharidin solution; Drug: Prednisolone; Drug: Placebo to prednisolone
- Cantharidin exposure to optimise blister formation (Experimental): Cantharidin exposure to optimise blister formation
  Interventions: Drug: Cantharidin solution

INTERVENTIONS:
Drug: Cantharidin solution — 5 microlitres of 0.025 to 0.5% topically on Day 1, 2 and 3
Drug: Aspirin — 300mg three times daily orally over a course of 4 days (starting Day -3) Part 2 only
  Arms: Effect of Aspirin
Drug: Prednisolone — 30mg orally once a day over a course of 4 days (starting Day -3) Part 2 only
  Arms: Effect of steroid - Prednisolone
Drug: Placebo to aspirin — 0mg three times daily orally over a course of 4 days (starting Day -3) Part 2 only
  Arms: Effect of Aspirin
Drug: Placebo to prednisolone — 0mg orally once a day over a course of 4 days (starting Day -3) Part 2 only
  Arms: Effect of steroid - Prednisolone

SUMMARY:
The purpose of this study is to refine the cantharidin-induced blister assay in healthy volunteers as a model of inflammatory disease. The study is an experimental trial in healthy volunteers in two parts; Part 1 to optimise the model and Part 2 to validate using two anti-inflammatory treatments with different modes of action.

DETAILED DESCRIPTION:
The purpose of this study is to refine the cantharidin-induced blister assay. The cantharidin-induced skin blister assay may be a valuable tool for evaluation of the pharmacodynamic effects of novel anti-inflammatory drugs in healthy volunteers, particularly for novel concepts targeting neutrophilic or monocytic inflammation. The study is an experimental trial in healthy volunteers for the purpose of evaluating the variability (between subjects and within subject) of the size and contents (cellular and fluid) of blisters induced on the forearm by direct application of cantharidin. Specifically, the aim is to assess whether variability is reduced in the current study, in which cantharidin will be applied directly to the skin in order to minimise the variation in total skin exposure. Once experimental design has been optimised then Part 2 of the study will examine the effects of a course of anti-inflammatory treatment prior to induction of blisters on the size and/or contents of blisters in a single blind crossover protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, vital signs, complete blood count and clinical chemistry. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Male between 18 and 55 years of age inclusive, at the time of signing the informed consent
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* Subjects with very fair or very dark skin type
* Presence on either forearm of tattoos, naevi, scars, keloids, hyperpigmentation, excessive hair or any skin abnormalities that may, in the opinion of the Investigator, interfere with study assessments
* Subjects with a history of keloids, skin allergy, hypersensitivity or contact dermatitis, including previous reactions to dressings to be used in the study
* Subjects with a history of lymphangitis and/or lymphoedema
* Subjects with a history of HIV infection, hepatitis B or C
* A positive pre-study drug/alcohol screen
* Use of prescription or non-prescription drugs, including ergot derivatives e.g. dihydroergotamine (Dihydergot), vitamins, herbal and dietary supplements (including St John's Wort) within whichever is the longer period of 7 days or 5 half-lives (if known) prior to the first challenge day, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56-day period For Part 2 only
* History of previous peptic ulcers, gastritis, GI bleed or history of bleeding problems, e.g. haemorrhoids or spontaneous nose bleeds
* Subjects with a history of asthma
* For aspirin only: History of sensitivity to aspirin or non steroidal anti-inflammatory drugs or a history of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor contraindicates their participation
* For prednisolone only: Subjects with systemic infections, hypersensitivity to any formulation ingredient, or ocular herpes simplex will be excluded. Those with, or a previous history of, tuberculosis, hypertension, congestive heart failure, liver failure, renal insufficiency, diabetes mellitus or in those with a family history of diabetes, osteoporosis, glaucoma or in those with a family history or glaucoma, subjects with a history of severe affective disorders and particularly those with a previous history of steroid-induced psychoses (in themselves or first degree relatives), epilepsy, peptic ulceration or previous steroid myopathy will also be excluded
* For prednisolone only: if a subject has not had chicken pox previously
* For prednisolone only: no live vaccines to be administered within 3 months of last prednisolone dose
* Subjects with a history of diabetes and peripheral vascular disease

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08-17 (Actual); Primary Completion 2011-01-14 (Actual); Study Completion 2011-01-14 (Actual)

PRIMARY OUTCOMES:
Blister volume of fluid | 48 hours
  Volume of fluid extracted from blisters induced by cantharidin application
Cell population in blister fluid | 48 hours
  Flow cytometry performed on cells from blister fluid including measurement of some or all of the following parameters: CD45, CD16, CD14, cell viability, CD206, CD64 or CD84, apoptosis, total blister leukocytes (CD45+), monocytes (CD14+), neutrophils (CD16 high), monocyte/macrophage like cells (CD64+ or CD84+); subsets of these cells that are undergoing apoptosis; subsets of monocyte/macrophages
Inflammatory mediators in blister fluid | 48 hours
  Inflammatory mediators in blister fluid, measured by immunoassay as primary endpoints may include (but will not be limited to): MPO, IL-10, IL-8, IL-6, IL-1β, TNF-α, LTB4.

SECONDARY OUTCOMES:
Blister volume of fluid | 72 hours
  Volume of fluid extracted from blisters induced by cantharidin application
Cell population in blister fluid | 72 hours
  Flow cytometry performed on cells from blister fluid including measurement of some or all of the following parameters: CD45, CD16, CD14, cell viability, CD206, CD64 or CD84, apoptosis, total blister leukocytes (CD45+), monocytes (CD14+), neutrophils (CD16 high), monocyte/macrophage like cells (CD64+ or CD84+); subsets of these cells that are undergoing apoptosis; subsets of monocyte/macrophages
Inflammatory mediators in blister fluid | 72 hours
  Inflammatory mediators in blister fluid, measured by immunoassay as primary endpoints may include (but will not be limited to): MPO, IL-10, IL-8, IL-6, IL-1β, TNF-α, LTB4.
Numbers and types of leukocytes in blood, and inflammatory mediators in plasma | 72 hours
Blister healing/skin appearance at 6 week follow up | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

REFERENCES:
- See also: Results for study 114416 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114416?search=study&search_terms=114416#rs